CLINICAL TRIAL: NCT01987622
Title: Acupuncture for Lumbar Spinal Stenosis: a Parallel, Randomized Controlled Pilot Study With Usual Care Comparison
Brief Title: Acupuncture for Lumbar Spinal Stenosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Korean Medicine Hospital of Pusan National University (Other)
Collaborators: Korea Institute of Oriental Medicine (Other Government)
Responsible Party: Principal Investigator, Gi Young Yang, Assistant Professor, Korean Medicine Hospital of Pusan National University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Acustenosis; KIOM (Other Grant/Funding Number: Korea Institute of Oriental Medicine)
Record Dates: First submitted 2013-11-12; First posted 2013-11-19 (Estimated); Last update posted 2015-02-09 (Estimated); Status verified 2015-02

CONDITIONS: Spinal Stenosis
Keywords: lumbar spinal stenosis; claudication; low back pain; radiculopathy; acupuncture; Korean medicine; randomized controlled trial
MeSH Terms: conditions — Spinal Stenosis; Intermittent Claudication; Low Back Pain; Radiculopathy | interventions — Acupuncture Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Acupuncture (Experimental): A series of acupuncture sessions within six weeks from the baseline
  Interventions: Procedure: Acupuncture; Procedure: Usual care
- Usual care (Active Comparator): An intervention consisting of patient education for a healthier lifestyle, including diet, exercise, self-management of symptoms, and the use of other treatments as needed.
  Interventions: Procedure: Usual care

INTERVENTIONS:
Procedure: Acupuncture — The patients in this group will receive individualized acupuncture prescribed by a certified Korean Medicine Doctor (KMD) with at least three years of clinical experience. The acupuncture formulas will be determined based on the individual patient's symptoms and at the KMD's discretion. The acupuncture treatment will be applied one to three times a week for six weeks (a total of 12 sessions and an additional four sessions are allowed). Acupuncture will be manually stimulated at first, and then electrical stimulation will be allowed at the KMD's discretion. Retention time will be equal to or less than 20 minutes. Examples of acupuncture points to be used might include LI4, LI11, TE5, SI3, TE3, ST36, SP6, SP9, LR3, GB34, Gb39, BL40, BL57, EX-B2, and BL23.
  Arms: Acupuncture
Procedure: Usual care — Usual care consists of patient education for a healthier lifestyle, including diet, exercise, self-management of symptoms, and the use of other treatments as needed. Participants will receive a three-page leaflet of patient education material. Optional regular physical therapies, including interferential current therapy (ICT) and local heat application, will be provided only for the control group at the participants' request . Physical therapy will be provided one to three times a week for six weeks (a total of 12 sessions and an additional four sessions are allowed). All kinds of conservative interventions for lumbar spinal stenosis, including analgesics and non-study physical treatments,will be allowed. However, surgical treatments, non-study acupuncture, or herbal medicine will not be allowed.

SUMMARY:
Acupuncture is widely used to manage chronic low back pain. Mounting evidence suggests the beneficial effects of acupuncture for mitigating chronic low back pain with acceptable minor adverse events. However, little information exists regarding the effects and safety of acupuncture for degenerative lumbar spinal stenosis, one of the spinal disorders that present chronic low back and leg pain.

The investigators aimed to assess the overall effectiveness, safety, and feasibility of acupuncture in combination with usual care (as opposed to usual care alone) for patients with symptomatic degenerative lumbar spinal stenosis.

The hypotheses of this study are as follows:

1. A set of acupuncture sessions in combination with usual care can provide greater functional improvements than usual care alone .
2. A set of acupuncture sessions in combination with usual care can provide greater pain reduction than usual care alone .

The study aims to include 50 participants (25 in the acupuncture group and 25 in the usual care group).

ELIGIBILITY:
Inclusion Criteria:

* Aged over 40
* Pain or bothersomeness of lower back or leg began at least three months ago (with at least 40 of pain or bothersomeness visual analogue intensity at the time of recruitment; 0 refers to no pain or bothersomeness and 100 to worst pain or bothersomeness imaginable)
* Clinical features of lumbar spinal stenosis, including neurological claudication or postural symptom changes
* Lumbar spinal stenosis confirmed by radiologic examination (e.g., computed tomography or magnetic resonance imaging) within the last two years
* Willingness to participate in the study

Exclusion Criteria:

* Congenital spinal stenosis
* Other spinal deformities, including spinal fractures and infections
* Participants who have received spinal surgeries, such as laminectomy, spinal fusion, and discectomy, due to lumbar spinal stenosis or other spinal diseases
* Other surgeries which might influence clinical features of lumbar spinal stenosis (e.g., total hip/knee replacements)
* Comorbid conditions which might interfere with the participant's active participation in the study (i.e., poorly controlled hypertension, poorly controlled diabetes mellitus, severe coronary artery disease, unstable asthma, cognitive function disorders, and other disabling conditions that interfere with self-ambulation, such as severe hip or knee arthritis)
* Past/present history of malignancy
* Began a new intervention for the management of lumbar spinal stenosis within the last one month
* Cauda equine syndrome (progressive lower extremity muscle weakness, loss of bowel/bladder control, and/or perianal numbness) and other urgent conditions which require immediate surgery
* Other conditions not appropriate for study participation

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2013-11; Primary Completion 2014-09 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Mid-term Back specific functional status | 3 months
  Participant-perceived reduction of pain and physical function will be measured with a 10-item questionnaire; change from baseline in the Oswestry Disability Index (ODI) scale will be used.

SECONDARY OUTCOMES:
Short-term Back specific functional status | 6 weeks
  Participant-perceived reduction of pain and physical function will be measured by a 10-item questionnaire; change from baseline in the Oswestry Disability Index (ODI) scale will be used.
Short-term low back pain bothersomeness | 6 weeks
  Participant-perceived reduction of bothersomeness due to low back pain will be measured by visual analogue scale (VAS) with range of 0 (no bothersomeness) to 100 (worst possible bothersomeness). Change from baseline in VAS scale will be used.
Mid-term low back pain bothersomeness | 3 weeks
  Participant-perceived reduction of bothersomeness due to low back pain will be measured by visual analogue scale (VAS) with range of 0 (no bothersomeness) to 100 (worst possible bothersomeness). Change from baseline in VAS scale will be used.
Short-term low back pain intensity | 6 weeks
  Participant-perceived reduction of low back pain intensity will be measured by visual analogue scale (VAS) with range of 0 (no pain) to 100 (worst possible pain). Change from baseline in VAS scale will be used.
Mid-term low back pain intensity | 3 weeks
  Participant-perceived reduction of low back pain intensity will be measured by visual analogue scale (VAS) with range of 0 (no pain) to 100 (worst possible pain). Change from baseline in VAS scale will be used.
Short-term leg pain bothersomeness | 6 weeks
  Participant-perceived reduction of bothersomeness due to radicular pain in leg will be measured by visual analogue scale (VAS) with range of 0 (no bothersomeness) to 100 (worst possible bothersomeness). Change from baseline in VAS scale will be used.
Mid-term leg pain bothersomeness | 3 months
  Participant-perceived reduction of bothersomeness due to radicular pain in leg will be measured by visual analogue scale (VAS) with range of 0 (no bothersomeness) to 100 (worst possible bothersomeness). Change from baseline in VAS scale will be used.
Short-term leg pain intensity | 6 weeks
  Participant-perceived reduction of leg pain intensity will be measured by visual analogue scale (VAS) with range of 0 (no pain) to 100 (worst possible pain). Change from baseline in VAS scale will be used.
Mid-term leg pain intensity | 3 months
  Participant-perceived reduction of leg pain intensity will be measured by visual analogue scale (VAS) with range of 0 (no pain) to 100 (worst possible pain). Change from baseline in VAS scale will be used.
Short-term pain-related quality of life | 6 weeks
  Patient-perceived improvement of pain-related quality of life will be measured by 2-item questionnaire for the subdomain of bodily pain in the Short-Form 36 Rand Health Insurance study batteries (SF-36) questionnaire. Change from baseline in bodily pain subdomain scale will be used.
Mid-term pain-related quality of life | 3 months
  Patient-perceived improvement of pain-related quality of life will be measured by 2-item questionnaire for the subdomain of bodily pain in the Short-Form 36 Rand Health Insurance study batteries (SF-36) questionnaire. Change from baseline in bodily pain subdomain scale will be used.
Short-term physical function-related quality of life | 6 weeks
  Patient-perceived improvement of physical function-related quality of life will be measured by 10-item questionnaire for the subdomain of physical function in the Short-Form 36 Rand Health Insurance study batteries (SF-36) questionnaire. Change from baseline in physical function subdomain scale will be used.
Mid-term physical function-related quality of life | 3 months
  Patient-perceived improvement of physical function-related quality of life will be measured by 10-item questionnaire for the subdomain of physical function in the Short-Form 36 Rand Health Insurance study batteries (SF-36) questionnaire. Change from baseline in physical function subdomain scale will be used.
Self-reported pain-free walking distance | 6 weeks, 3 months
  Patient-reported pain-free walking distance with providing the actual reference distance of 50 meters in the corridor of the research center.
Patient satisfaction for treatment outcome | 6 weeks, 3 months
  Patients' satisfaction for allocated treatment outcomes will be measured by a single item with 7-point likert scale question (very much satisfied, much satisfied, a bit satisfied, just the same, a bit dissatisfied, much dissatisfied, very much dissatisfied).
Patient Global Assessment for treatment outcome | 6 weeks, 3 months
  Patients' global assessment for overall treatment outcome will be measured by a single item with 5-point likert scale question (much improved, somewhat improved, just the same as baseline, somewhat worsened, much worsened)
Use of medication and healthcare resources | 6 weeks, 3 months
  Information on the use of medication and other non-study healthcare resources will be collected by directly asking the patient at every visit. Patients in the control group who do not visit the research center to receive optional physical therapies will be contacted regularly by short-form message service and phone calling by study investigators. Examples of healthcare resources include analgesics, physical therapies, epidural injection, hospital visits for symptoms of lumbar spinal stenosis. Types and frequency of the use of healthcare resources will be assessed at 6 weeks and 3 months from baseline.
Adverse events | 6 weeks, 3 months
  All expected or unexpected adverse events in both groups will be measured at the every study visit as well as by the telephone interview. Types and frequency of the occurrence of adverse events will be assessed at 6 weeks and 3 months from baseline.

OTHER OUTCOMES:
Participant expectancy for allocated treatments | Baseline, 6 weeks, 3 months
  Each participant's expectancy for allocated treatment to reduce symptoms of lumbar spinal stenosis will be measured by a single-item questionnaire ("Do you think your allocated treatment will be [was] helpful to reduce your symptoms related to lumbar spinal stenosis?"). Possible answers will be 0 (not at all helpful) to 6 (very helpful).

CONTACTS AND LOCATIONS:
Overall Officials: Gi Young Yang, PhD, Principal Investigator — Korean Medicine Hospital, Pusan National University
Locations (1):
- National Clinical Research Center, Korean Medicine Hospital, Pusan National University, Yangsan, Kyungsangnamdo, South Korea

REFERENCES:
- [Derived] Kim KH, Kim YR, Baik SK, Noh SH, Kim DH, Lee SW, Yang GY. Acupuncture for patients with lumbar spinal stenosis: a randomised pilot trial. Acupunct Med. 2016 Aug;34(4):267-74. doi: 10.1136/acupmed-2015-010962. Epub 2016 Mar 7. PMID 26953235